CLINICAL TRIAL: NCT06350019
Title: Vascular hemodynamıc Effects of penılle revascularızatıon Surgery and the Role of resıstıve ındex ın Follow-up
Brief Title: Vascular Effects of Penil revascularızatıon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Fatih Akdemir, Assist. Prof., Ankara Yildirim Beyazıt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26379996/91
Record Dates: First submitted 2024-03-25; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Erectile Dysfunction; Erectile Dysfunction Due to Arterial Disease; Erectile Dysfunction Due to Venous Disorder
Keywords: Erectile dysfunction; Penile revascularization; Penile color doppler ultrasonography; Resistive index
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cases with erectile dysfunction of vascular origin (Experimental): Penile revascularization surgery was performed in cases with erectile dysfunction of vascular origin. Penile color Doppler ultrasonography, corpus cavernosum electromyography and cavernosometry tests were performed on all cases in the preoperative period and at the 3rd postoperative month. Penile computed tomography angiography was performed at the 3rd postoperative month.
  Interventions: Procedure: Penile revascularızation

INTERVENTIONS:
Procedure: Penile revascularızation — The importance of resistive index in the preoperative evaluation of vascular-induced erectile dysfunction, predicting the success of penile revascularization surgery, and postoperative patient management was investigated.

SUMMARY:
Purpose: The aim of this study is to measure the effects of penile revascularization surgery performed in vascular origin erectile dysfunction (ED) on penile vascular hemodynamic and to determine the importance of vascular parameters in postoperative patient follow-up.

Methods: A total of 35 participants who underwent penile revascularization surgery due to vascular ED were included in this study. In the preoperative period and at the 3rd postoperative month, penile color doppler ultrasonography (PCDU) was performed to evaluate cavernosal arteries, dorsal arteries, deep dorsal vein and inferior epigastric artery (IEA) separately. During this evaluation, peak systolic velocity (PSV), end diastolic velocity (EDV), and resistive index (RI) were measured. The International Index of Erectile Function questionnaire (IIEF) was applied to all patients in the preoperative period and at the 3rd postoperative month. The relationship between changes in (IIEF) questionnaire score and penile vascular hemodynamic changes in the postoperative period was evaluated.

DETAILED DESCRIPTION:
A total of 35 participants who underwent penile revascularization surgery with the diagnosis of vascular ED in our clinic were included in this study. Detailed anamnesis of the cases was taken, including age, duration of ED, comorbidities that may cause ED, previous trauma, medical or surgical history and lifestyle. After the physical examination, IIEF 5/15 questionnaires were filled out. In order to exclude hypogonadism, follicle stimulating hormone(FSH), luteinizing hormone(LH), total testosterone and prolactin levels were measured in the preoperative period. PCDU, CC-EMG and cavernosometry tests were applied to all participants in the preoperative period. Participants that did not benefit from phosphodiesterase 5 inhibitors(PDE-5I) and intracavernosal alprostadil injection used in the preoperative period were included in the study. Cases with a history of urogenital, rectal and similar operations that may affect erectile functions, cases with penile pathologies such as Peyronie's disease, and cases with ED of neurogenic and psychogenic origin were excluded from this study. After the 3rd postoperative month, participants were interviewed face to face. During these follow up, the patients were re-evaluated with the IIEF-5/15 questionnaires, and PCDU and computurized tomography angiography (CTA) was performed.

PCDU technique: The PCDU was performed in a quiet and comfortable room for the participants' comfort. For the diagnosis of arterial insufficiency or veno-occlusive disease, PCDU(B-K Medical, Herlev, Denmark) was performed with the patient lying in the supine position. First, gray scale imaging of the flaccid penil shaft in transverse and sagittal planes was performed to exclude intracavernosal fibrosis and calcifications. Then, 60 mg papaverine hydrochloride (Papaverine HCl®, Galen Medical Industry, Turkey) was injected laterally into any of the corpus cavernosum with a 22 Gauge needle. 20 minutes after papaverine HCl injection, PCDU was performed with an 8 Megahertz (MHz) linear probe at an angle of approximately 45 degrees. PSV, EDV, RI values of both cavernosal arteries and anastomosis region were calculated. Measurements were repeated at 5-minute intervals and continued for 30 minutes. Participants with PSV<25 cantimeters/second (cm/s) were interpreted as arterial insufficiency, and participants with PSV>25 cm/s, EDV >5 cm/s and RI<0.85 were interpreted as veno-occlusive disease. RI was calculated with the formula [RI=(PSV-EDV)/PSV]. Participants were warned about the risk of priapism after papaverine HCl injection and were asked to immediately consult the clinic if the erection persisted after four hours.

CC-EMG technique: Penil cavernous electrical activity (CEA) was recorded using a high-speed electromyography module equipped with a computer (Medical Measurement Systems, Enschede, the Netherlands). The sampling frequency was 200 Hertz (Hz), and a band-pass ﬁlter with a cut-off frequency of 0.1-20 Hz was used. During the CC-EMG recordings, monopolar needle electrode was used to measure the CEA. A grounding electrode was placed to the participants' foot to avoid electrical activity simultaneously originating from non-penil areas. It appears as a single line in the CC-EMG recording. CC-EMG recordings were started after the participants rested for 10 minutes in a quiet and dim room. CEA potentials were recorded for 10 minutes. Later the CEA potentials of the penil cavernous nerves was assessed by detecting the peak-to-peak amplitudes. Ten minutes later, papaverine HCl (60 mg) was injected into a single cavernous body for avoiding the pattern of discoordination, which manifested by an increase or no difference in the CEA recording following the injection and suggested the neurogenic ED. Participants with a discoordination pattern were not included in the study. The relaxation degree (RD) was calculated using the formula: RD=Pre-injection CEA-Post-injection CEA/Preinjection CEA×100, as previously described. Participants having less than 50% RD were excluded from the study.

Cavernosometry technique: After CC-EMG recordings were made, cavernosometry was conducted with the same device. In the presence of the following criteria, a diagnosis of caverno-occlusive dysfunction was made.

1. Requires a maintenance flow rate greater than 5 milliliters/minute (ml/m) after revealed an intracavernous pressure of 150 millimeters-Hg (mmHg) with the artificial erection test.
2. The intracavernous pressure decreased by a minimum of 45 mmHg within 30 second following the termination of infusion.

Surgical technique: The operations, were conducted using the Furlow-Fisher procedur, of the Virag-V technique. Unlike the Furlow- Fisher procedure, the circumﬂex collaterals were preserved, and the deep dorsal venous valves were not disrupted by a stripper. After the IEA was brought to the penil root through the subcutaneous tunnel, an end-to-side anastomosis was performed with the proximal part of the deep dorsal vein. 7-0 polypropylene suture were used according to a standard microsurgical procedure. After the anastomosis, the deep dorsal vein was ligated proximal to the arteriovenous anastomosis. The procedure was performed under optical magnification (x2.5) to prevent neurovascular bundle damage. In the postoperative period, intravenous heparin (5000 IU/day) was prescribed for 3 days, 75 mg/day dipyridamole and 300 mg/day acetylsalicylic acid daily for three months. He was warned not to have sexual intercourse for 2 months after the operation.

CTA technique: In the third postoperative month, participants underwent CTA. 60 milligram (mg) papaverine HCl was administered to the subjects 10 minutes before the shooting. A 22-gauge branule was placed in the basilic or cephalic vein of the patient's forearm. Then, the patient was placed supine on the imaging stretcher and the area to be imaged was determined. Then, using an automatic injector pump, iodinated contrast material(Iopromide, Ultravist®, Schering, Germany) was given to the patient intravenously at a dose of 2 mg/kg and at a flow rate of 3 ml/s. Then, arterial phase pelvic CTA with 2 mm slice thickness was performed with a 64-detector, multi detector CT machine (Aquilion 64, Toshiba®, Tokyo, Japan). After CTA examination, sagittal and coronal reformatted images(slice thickness: 1 mm) were obtained. CT images were evaluated by an experienced radiologist.

ELIGIBILITY:
Inclusion Criteria:

* Cases that do not benefit from oral phosphodiesterase 5 inhibitor or intracavernosal injection treatment
* Cases with PSV<25 cm/s in PCDU
* Cases with PSV>25 cm/s, EDV>5 cm/s and RI<0.85 in PCDU
* Patients with relaxation degree above 50% in CC-EMG
* Cases with venous leakage in cavernosometry

Exclusion Criteria:

* hypogonadism (primer or secondary),
* Cases benefiting from phosphodiesterase 5 inhibitors
* Cases benefiting from intracavernous alprostadil
* Those with a history of urogenital, rectal and similar operations
* Those with Peyronie's disease
* Cases of neurogenic and psychogenic origin

Ages: 23 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All cases included in the study were male individuals.
Enrollment: 35 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-08-15 (Actual); Study Completion 2014-12-25 (Actual)

PRIMARY OUTCOMES:
The importance of resistive index in evaluating the postoperative success of penile revascularization | 3 months (Postoperative third months)
  Penile revascularization was performed in 35 cases with the diagnosis of erectile dysfunction of vascular origin. Both preoperative and postoperative international index of erectile function questionaire (IIEF) and penile color Doppler ultrasound (PCDU) were performed in all cases, and IIEF 5/15 scores and resistive index (RI) were calculated. After the operation, computerized tomography angiography (CTA) was performed to confirm anastomotic patency. The correlation between RI and IIEF was evaluated in the postoperative period. RI = 0.85 was accepted as the limit value to evaluate postoperative success. Cases with RI>0.85 were considered successful and cases with RI<0.85 were considered unsuccessful.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih AKDEMİR, Principal Investigator — Ankara Yildirim Beyazıt University

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available

REFERENCES:
- [Derived] Akdemir F, Kayigil O. Vascular hemodynamic effects of penile revascularization surgery and the role of resistive index in follow-up. Basic Clin Androl. 2024 Dec 20;34(1):28. doi: 10.1186/s12610-024-00243-0. PMID 39701967